CLINICAL TRIAL: NCT04375098
Title: Efficacy and Safety of Early Anti-SARS-COV-2 Convalescent Plasma in Patients Admitted for COVID-19 Infection: a Randomized Phase II Trial
Brief Title: Efficacy and Safety of Early COVID-19 Convalescent Plasma in Patients Admitted for COVID-19 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Fundacion Arturo Lopez Perez (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200415015
Record Dates: First submitted 2020-05-03; First posted 2020-05-05 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2
Keywords: Plasma; COVID-19; severe acute respiratory syndrome coronavirus 2
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early COVID-19 convalescent plasma (Experimental): COVID-19 convalescent plasma 200 ml day 1 and 2 at admission after confirmation of eligibility
  Interventions: Biological: COVID-19 convalescent plasma
- COVID-19 convalescent plasma (Experimental): COVID-19 convalescent plasma 200 ml day 1 and 2 only if worsening of respiratory function or persistence of COVID symptoms for >7 days after enrolment
  Interventions: Biological: COVID-19 convalescent plasma

INTERVENTIONS:
Biological: COVID-19 convalescent plasma — COVID-19 convalescent plasma

SUMMARY:
Currently there is no standard treatment for SARS-CoV-2 infection. Use of convalescent plasma has been studied in outbreaks of other respiratory infections, including SARS-CoV-1 , MERS-CoV and Hantavirus infection. This study is an open-label randomized trial in which patients with high risk of COVID19-associated respiratory failure will be randomized to early treatment with convalescent plasma (≤ 7 days from symptoms start) or at early signs of respiratory failure or prolonged hospitalization. COVID-19 convalescent plasma will be collected from individuals according to the institutional protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years
* CALL score ≥ 9 (progression risk score)
* PCR-confirmed COVID-19 infection with equal or less than 7 days of symptoms (or imaging consistent with COVID-19 pneumonia and confirmed COVID-19 contact)
* Any symptoms of COVID-19 infection
* Admission due to COVID-19 infection
* Signed informed consent
* ECOG before COVID-19 infection 0-2

Exclusion Criteria:

* PaFi <200 or mechanical ventilation indication
* Clinically relevant co-infection at admission
* Pregnancy or lactation
* IgA deficiency or IgA nephropathy
* Immunoglobulin or plasma administration in the last 60 days
* Contraindication to transfusion or previous allergy to blood-derived products
* Do-not-resuscitate status
* Patients receiving other investigational drug for COVID-19 in a clinical trial
* Any condition, that in opinion of the investigator may increase the risk associated with study participation or interfere with the interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Percentage Mechanical Ventilation, hospitalization longer than 14 days or death during hospitalization | 1 year follow up

SECONDARY OUTCOMES:
Median duration of fever | 1 year
  Days
Median duration of mechanical ventilation | 1 year follow up
  Days
Median length of ICU stay | 1 year follow up
  Days
Median length of admission | 1 year follow up
  Days
Hospital mortality rate (percentage) | 1 year follow up
30-day mortality (percentage) | 1 year follow up
Readmission rate (percentage) | 1 year follow up
Median length of viral clearance | 1 year follow up
  days

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elvira Balcells, MD, Principal Investigator — ebalcells@uc.cl
Locations (1):
- Hospital Clínico Universidad Católica, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Gharbharan A, GeurtsvanKessel CH, Jordans CCE, Blaauw M, van der Klift M, Hassing RJ, Smits-Zwinkels M, Meertens M, van den Hout EC, de Man AM, Hageman I, Bogers S, van der Schoot CE, Swaneveld F, Anas AA, Rokx C, Rijnders BJA. Effects of Treatment of Coronavirus Disease 2019 With Convalescent Plasma in 25 B-Cell-Depleted Patients. Clin Infect Dis. 2022 Apr 9;74(7):1271-1274. doi: 10.1093/cid/ciab647. PMID 34293119
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969
- [Derived] Balcells ME, Rojas L, Le Corre N, Martinez-Valdebenito C, Ceballos ME, Ferres M, Chang M, Vizcaya C, Mondaca S, Huete A, Castro R, Sarmiento M, Villarroel L, Pizarro A, Ross P, Santander J, Lara B, Ferrada M, Vargas-Salas S, Beltran-Pavez C, Soto-Rifo R, Valiente-Echeverria F, Caglevic C, Mahave M, Selman C, Gazitua R, Briones JL, Villarroel-Espindola F, Balmaceda C, Espinoza MA, Pereira J, Nervi B. Early versus deferred anti-SARS-CoV-2 convalescent plasma in patients admitted for COVID-19: A randomized phase II clinical trial. PLoS Med. 2021 Mar 3;18(3):e1003415. doi: 10.1371/journal.pmed.1003415. eCollection 2021 Mar. PMID 33657114